CLINICAL TRIAL: NCT00533013
Title: Comprehensive Program for Disease Management in Heart Failure Patients in the Community
Brief Title: Comprehensive Heart Failure Disease Management Community Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Ofra Kalter-Leibovici MD, Dr. Ofra Kalter-Leibovici, Maccabi Healthcare Services, Israel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-07-4807-OK-CTIL
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Disease Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Management of heart failure is provided by primary practitioners and consultant cardiologists
  Interventions: Other: Usual Care
- Disease Management (Experimental): Disease management led by nurse specialists in regional Heart Failure Clinics and a national Call Center. Tele-Monitoring of body weight, pulse rate and blood pressure is performed at participants' homes.
  Interventions: Other: Disease Management and Tele-Monitoring

INTERVENTIONS:
Other: Usual Care — Management of heart failure is provided by primary practitioners and consultant cardiologists
  Arms: Usual care
Other: Disease Management and Tele-Monitoring — Management of heart failure is provided by cardiologists at regional heart failure clinics and by nurse practitioners at regional heart failure clinics and a designated call center. Decisions on treatment are guided by designated protocols and information derived for tele-monitoring of blood pressure, body weight and pulse rate.
  Arms: Disease Management

SUMMARY:
The purpose of this study is to determine whether a nurse-led, comprehensive disease management program is effective in reducing recurrent hospital admissions and deaths in community dwelling patients with moderate to severe heart failure.

DETAILED DESCRIPTION:
Heart failure remains a significant cause of death, in spite of recent declines in overall mortality from cardiovascular disease. Heart failure is associated with increasing costs for healthcare, mainly for recurrent hospital admissions. Disease management programs aimed to improve patients outcome while containing healthcare costs,were employed in heart failure patients with varying results. Such programs contain various components, including patient education and empowerment, monitoring patients' adherence to therapy, telemonitoring of vital parameters, etc. Designated heart failure clinics were also employed in care given to these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with NYHA-Stage III-IV heart failure recruited in the community;
2. Adult patients with NYHA-Stage II-IV heart failure recruited after hospital admission for decompensated heart failure

Exclusion Criteria:

* Other severe disease (e.g. end stage renal disease, metastatic cancer); bedridden or severely compromised functional status due to other diseases; drug or alcohol abuse; Severe cognitive impairment; People unconnected to telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1360 (Actual)
Dates: Start 2007-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
hospital admissions for heart failure or all-cause mortality | 5 years

SECONDARY OUTCOMES:
Health-related Quality of Life; | 5 years
  SF-36 score
Functional status | 5 years
  6-minute walk-test; NYHA classification category

CONTACTS AND LOCATIONS:
Overall Officials: Haim Silber, M.D., Principal Investigator — Maccabi Healthcare Services, Israel; Ofra Kalter-Leibovici, M.D., Principal Investigator — Sheba Medical Center; Galit Kaufman, RN, Study Director — Sheba Medical Center
Locations (1):
- Maccabi Health Services, Tel Aviv, Israel

REFERENCES:
- [Result] Kalter-Leibovici O, Freimark D, Freedman LS, Kaufman G, Ziv A, Murad H, Benderly M, Silverman BG, Friedman N, Cukierman-Yaffe T, Asher E, Grupper A, Goldman D, Amitai M, Matetzky S, Shani M, Silber H; Israel Heart Failure Disease Management Study (IHF-DMS) investigators. Disease management in the treatment of patients with chronic heart failure who have universal access to health care: a randomized controlled trial. BMC Med. 2017 May 1;15(1):90. doi: 10.1186/s12916-017-0855-z. PMID 28457231
- [Derived] Kalter-Leibovici O, Murad H, Ziv A, Keidan T, Orion A, Afel Y, Gilutz H, Freimark D, Klibansky-Marom R, Freedman L, Silber H. Causes and predictors of recurrent unplanned hospital admissions in heart failure patients: a cohort study. Intern Emerg Med. 2024 Nov;19(8):2213-2221. doi: 10.1007/s11739-024-03740-2. Epub 2024 Aug 18. PMID 39154298